CLINICAL TRIAL: NCT05232747
Title: Determination of Behavioral and Emotional Factors Associated With Pain Severity in Patients With Chronic Low Back Pain
Brief Title: Behavioral and Emotional Factors Associated With Pain Severity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Principal Investigator, Suleyman Demirel University
Other Study IDs: 72867572-050.01.04-196254
Record Dates: First submitted 2022-01-28; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Back pain; Pain Beliefs; Pain Coping; Behavioral; Emotional
MeSH Terms: conditions — Back Pain; Behavior | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study: Participants' pain level and pain-related behaviors will be questioned.
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Diagnostic Test

SUMMARY:
The planned research will address the behavioral and emotional factors associated with low back pain rather than a structural and biological cause. It will be determined to what extent the results obtained according to the ICF model are effective on the participation of patients with low back pain in daily activities, and it will become clear whether patients with low back pain should be approached only mechanically in the rehabilitation programs.

DETAILED DESCRIPTION:
Chronic low back pain is among the most important health and economic problems of today. In particular, the success of chronic low back pain treatment with current approaches based on the biomedical care model, which is thought to be synonymous with pain and tissue damage, is limited. It has been demonstrated that tissue damage is not a prerequisite for the development of chronic low back pain. Several studies have shown a strong association between chronic low back pain and psychological factors such as anxiety, fear avoidance, distress/depressed mood, anger, poor coping strategies, and low pain self-efficacy. Despite all this important information and evidence, there is a lack of an overview of the behavioral and emotional factors associated with pain severity, as studies mostly focus on a few major factors. However, the strong interaction between behavioral and emotional factors leads to confusion.

The psychological factors mentioned above are open to discussion, and people with chronic low back pain may experience increased pain severity as a result of emotional processing inadequacy. Baker et al identified five factors for emotional processing deficits related to emotion suppression, unprocessed emotion symptoms, unregulated emotion, avoidance, and poor emotional experience. It is hypothesized that the stated emotional processing deficits have a potential role in the increase in pain severity and development of pain in individuals with chronic low back pain. Therefore, depending on the severity of emotional processing openness, the person may feel pain more than it actually is, exhibit more fear avoidance behavior, and develop negative coping strategies with pain. More recently, Baker et al. argued that the sensation of pain lies at the interface between physical and psychological processes, and therefore, impaired emotional processing may be associated with both psychological factors and physical conditions such as chronic low back pain. However, it is currently unknown whether patients with chronic low back pain process pain sensation differently from asymptomatic individuals. Therefore, behavioral and emotional factors related to pain severity have not been clearly revealed.

The aim of this study is to determine the behavioral and emotional factors associated with pain severity in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-55 years old
* Having a history of chronic low back pain for at least 3 months
* Having a low back pain level of 1 or higher according to the Visual Analog Scale

Exclusion Criteria:

* Having had any surgery on the lumbar region
* Having a history of lower extremity surgery
* Having acute low back pain
* Having a neurological disease
* Having sensory loss
* Presence of a rheumatological disease that may cause low back pain
* Having a herniated disc pressing on the sacral nerves
* being pregnant

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with low back pain
Sampling Method: Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Visuel Analog Scale | 3 months
  Visual Analogue Scale will be used to evaluate the severity of low back pain. The back pain they feel during activity and rest will be questioned separately from the participants. For this assessment, patients will be asked to mark their pain intensity on a 10-centimeter line. Pain intensity will be determined by measuring the distance of the marked point to the "0" point with a tape measure. Scoring is done on a scale of 0-10 and "0 means no pain"- "10 means the most severe pain imaginable".
The Pain Beliefs Questionnaire | 3 months
  It was developed by Edwards et al. in 1992 to evaluate beliefs about the cause and treatment of pain. In our country, the validity and reliability study of the scale was carried out by Berk in 2006 and it was adapted to Turkish. There are 12 items in this scale covering pain beliefs. Accordingly, the scale consisted of two test areas: Organic Beliefs consisting of 8 items and Psychological Beliefs consisting of 4 items. The Organic Belief test reflects that the pain is largely of organic origin. (For example, 'pain is caused by damage to tissues in the body' and 'pain experience is a sign of something wrong with the body.) Psychological Belief test shows that the experience of pain is under the influence of psychological factors. (For example, 'worrying makes the pain worse.' 'thinking about the pain makes the pain worse').
Pain Coping Questionnaire | 3 months
  It was developed by Kleinke in 1992 to reveal pain-specific affect and behavior patterns. The scale assesses the way chronic pain patients cope with organic or psychogenic pain. The validity and reliability study of the scale was performed by Karaca et al. in 1996 and adapted to Turkish. The scale consists of 4 subtests. These; Self-Coping, Helplessness, Conscious Cognitive Interventions, Medical Remedy Seeking subtests.
Fear-Avoidance Beliefs Questionnaire | 3 months
  It has 16 questions and two subscales: physical activity and work. The physical activity section consists of 5 questions and the labor section consists of 11 questions. The questionnaire is a 7-point Likert type scale. In the answers given to the questionnaire, 0 points are given to the statement of "I don't agree at all" and 6 points to the statement of "I totally agree". Both subscale scores can be used independently. There are 16 questions in the original of the CCSI developed by Waddell. It is accepted that there is a decrease in fear-avoidance behavior within the department as the total score approaches 0 in the evaluation, and an increase in fear-avoidance behavior as it approaches the maximum score.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Duray, Principal Investigator — Suleyman Demirel University
Locations (1):
- Mehmet Duray, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No